CLINICAL TRIAL: NCT00695032
Title: Biologic Evaluation of Renal Toxicity of Cisplatin and Ifosfamide (TOXIPLAT)
Brief Title: Kidney Damage in Patients Receiving Cisplatin and Ifosfamide for Solid Tumors
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 07GENE03; ICREGAUD-TOXIPLAT; ICREGAUD-07-GENE-03; EUDRACT-2007-004251-12; INCA-RECF0479
Record Dates: First submitted 2008-06-07; First posted 2008-06-11 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Chemotherapeutic Agent Toxicity; Renal Toxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: renal toxicity; chemotherapeutic agent toxicity; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cisplatin
Drug: ifosfamide
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and urine from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is evaluating kidney damage in patients receiving cisplatin and ifosfamide for solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify and evaluate the early biomarkers of renal toxicity in patients with solid tumors treated with cisplatin and ifosfamide.

Secondary

* Correlate the modification of biomarker studies and blood concentrations of cisplatin.

OUTLINE: Patients receive standard chemotherapy comprising cisplatin and/or ifosfamide.

Blood and urine samples are collected on days 1 and 2 (or day 3 if receiving ifosfamide only) during the first 3 courses. Samples are analyzed to determine plasma concentrations of residual cisplatin and to obtain urinary-protein profiles to measure renal toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a solid tumor

  * Any location allowed
  * Metastatic disease allowed
* Planned treatment comprising cisplatin and/or ifosfamide as standard chemotherapy

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Life expectancy > 3 months
* Creatinine clearance ≥ 60 mL/min
* Must be available for follow up
* Not pregnant or nursing
* Not under guardianship or in prison

Exclusion criteria:

* Prior drug-related nephrotoxicity
* Acute, uncontrolled urinary infection or > 48-hours
* Pre-existing hemorrhagic cystitis
* Weak bladder
* Bilateral obstruction of urinary tract
* Insufficient, severe bone marrow hypoplasia
* Cardiorespiratory condition contraindicating hyperhydration
* Hearing impairment
* Hypersensitivity to cisplatin or products containing platinum
* Major psychiatric condition (severe depression, psychosis, dementia)

PRIOR CONCURRENT THERAPY:

* No prior yellow fever vaccine, live attenuated vaccine, or phenytoin
* No concurrent participation in another biomedical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evolution of different biomarkers
Sensitivity, specificity, and predictive value (positive and negative) of different markers

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chevreau-Dalbianco, MD, Study Chair — Institut Claudius Regaud
Locations (1):
- Institut Claudius Regaud, Toulouse, France